CLINICAL TRIAL: NCT00268528
Title: Understanding the Ethnic and Racial Differences in Survival in Children With Acute Lymphoblastic Leukemia
Brief Title: Study to Assess Compliance With Long-Term Mercaptopurine Treatment in Young Patients With Acute Lymphoblastic Leukemia in Remission
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL03N1; NCI-2009-00305 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000459748; 07-462; AALL03N1 (Other: Childrens Oncology Group); COG-AALL03N1 (Other: DCP); AALL03N1 (Other: CTEP); R01CA096670 (NIH); U10CA095861 (NIH)
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2019-10

CONDITIONS: Childhood Acute Lymphoblastic Leukemia in Remission
MeSH Terms: interventions — Mercaptopurine; azathiopurine; Methotrexate; merphos

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health service research (electronic pill monitoring system): Patients receive an electronic pill monitoring system comprising an empty MEMS^? medication bottle with TrackCap? CR. The mercaptopurine prescription is filled using this system. Beginning on day 1 of the third or later course of maintenance therapy, patients take all doses of mercaptopurine from the MEMS^? medication bottle with TrackCap? CR for at least 169 days. The MEMS^? TrackCap? CR is mailed to the Coordinating Center at the end of study. Patients also receive methotrexate PO as indicated by their individual chemotherapy regimen.
  Interventions: Behavioral: Compliance Monitoring; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Other: Questionnaire Administration; Other: Study of Socioeconomic and Demographic Variables

INTERVENTIONS:
Behavioral: Compliance Monitoring — Receive an electronic pill monitoring system comprising an empty MEMS medication bottle with TrackCap
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; BW 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Other: Questionnaire Administration — Ancillary studies
Other: Study of Socioeconomic and Demographic Variables — Receive an electronic pill monitoring system comprising an empty MEMS medication bottle with TrackCap

SUMMARY:
This clinical trial is assessing compliance with long-term mercaptopurine treatment in young patients with acute lymphoblastic leukemia in remission. Assessing why young patients who have acute lymphoblastic leukemia may not take their medications as prescribed may help identify ways to assist them in taking their medications more consistently and may improve long-term treatment outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine and compare adherence to maintenance mercaptopurine (6-MP) in a cohort of children with acute lymphoblastic leukemia (ALL) from four different ethnic and racial groups (Caucasians, African-Americans, Hispanics, and Asians) receiving maintenance/continuation chemotherapy, using the following assessments: serial red cell 6-MP metabolites (6-thioguanine [6TGN] and methyl thioinosine monophosphate [TIMP]); frequency of 6-MP dosing using an electronic pill monitoring system (Microelectromechanical Systems [MEMS]?); self-report of adherence to 6-MP by questionnaire.

II. To determine the impact of adherence to 6-MP (measured using 6TGN, methyl [Me]TIMP, MEMS? and self-report data independently) on event-free-survival (EFS) in the entire cohort, after adjusting for known predictors of disease outcome.

III. Define a critical level of adherence (measured independently by 6TGN, MeTIMP, MEMS?, self-report) that has a significant impact on EFS for the entire cohort.

IV. Describe prevalence of adherence to 6-MP by ethnicity (6TGN, MeTIMP, MEMS?, Self-report).

V. Describe behavioral and socio-demographic predictors of adherence using the questionnaire data.

VI. Describe the pill-taking practices in this cohort using the MEMS? data. VII. To evaluate the impact of adherence on ethnic/racial difference in EFS.

SECONDARY OBJECTIVES:

I. To assess the concordance among 6TGN and MeTIMP levels, electronic pill monitoring, and self-reported adherence in the ethnic/racial groups.

OUTLINE:

Patients receive an electronic pill monitoring system comprising an empty MEMS? medication bottle with TrackCap? child resistant (CR). The mercaptopurine prescription is filled using this system. Beginning on day 1 of the third or later course of maintenance therapy, patients take all doses of mercaptopurine from the MEMS? medication bottle with TrackCap? CR for at least 169 days. The MEMS? TrackCap? CR is mailed to the Coordinating Center at the end of study. Patients also receive methotrexate orally (PO) as indicated by their individual chemotherapy regimen.

NOTE: *Study closed to accrual for Caucasian and Hispanic patients as of 8/14/2009.

After completion of study, patients are followed up every 6 months for 5 years and then annually for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALL in first remission, irrespective of risk stratification; enrollment on a Children's Oncology Group (COG) therapeutic study for ALL is not required, but the treatment plan must meet the criteria in this protocol
* Belongs to one of the four following ethnic/racial categories: African-American, Asian, Caucasian, or Hispanic; below please find definitions for these categories

  * African-American: includes patients who are African-American or of sub-Saharan black African ancestry
  * Asian: patients of Asian ancestry, including the following: Asian Indian (subcontinent), Chinese, Japanese, Korean, Native Hawaiian, Guamanian or Chamorro, Pacific Islander, Filipino, Vietnamese, Samoan, Hmong, Cambodian, Thai, Laotian, or Other Asian races
  * Caucasian: includes White or light-skinned patients of European, North African, or Middle Eastern ancestry
  * Hispanic: patients of Hispanic ethnicity, including the following: Mexican, Mexican American, Chicano, Cuban, Puerto Rican, or Other Spanish/Hispanic/Latino ethnicity
* Receiving self- or parent/caregiver-administered oral anti-metabolite chemotherapy during the maintenance/continuation phase of therapy; patients are eligible if their treatment plan calls for the following doses of 6-MP and methotrexate (MTX) during the maintenance/continuation phase: 6-MP ? 75 mg/m^2/day orally; MTX 20 mg/m^2/week orally;** (modification of 6-MP or MTX dosing based on laboratory or clinical parameters is acceptable)

  * For guidance regarding if and when a patient being treated on or according to a specific COG (or legacy group) protocol is eligible, please refer to ?AALL03N1 Eligibility by Protocol Tool,? available in the study data forms packet on the COG website
* Has completed at least 24 weeks of maintenance/continuation chemotherapy, and is scheduled to receive at least 24 more weeks of maintenance/continuation chemotherapy**

  * For guidance regarding if and when a patient being treated on or according to a specific COG (or legacy group) protocol is eligible, please refer to ?AALL03N1 Eligibility by Protocol Tool,? available in the study data forms packet on the COG website
* Written informed consent from the patient and/or the patient?s legally authorized guardian, obtained prior to registration and any study-related procedures, and in accordance with institutional policies approved by the United States (U.S) Department of Health and Human Services

Exclusion Criteria:

* Patients of multi-ethnic/multi-racial backgrounds are not eligible for this study; while patients of multi-ethnic/multi-racial ancestry (e.g., Caucasian/Japanese, Hawaiian/Puerto Rican) are not eligible, patients of mixed ancestry within a race/ethnicity (e.g., Japanese/Chinese = Asian or Korean/Japanese/Hawaiian = Asian or Mexican/Puerto Rican = Hispanic) may participate as long as they fall under the general classification of "African-American," "Asian," "Caucasian," or "Hispanic"

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with ALL from four different ethnic and racial groups (Caucasians, African-Americans, Hispanics, and Asians) receiving maintenance/continuation chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2005-05-30 (Actual); Primary Completion 2012-03-05 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to 6-MP as measured by 6TGN and MethylTIMP levels | 169 days
  Will initially perform an exploratory data analysis on distributions across the four groups using side-by-side boxplots, histograms, and summary quantities (mean, median, quartiles, standard deviations, inter-quartile-range, etc.). If central values summarize across-group differences well, then mean and median of the distribution will be compared between 6 pairs of the four ethnic groups using the two-sample t-test and the Mann-Whitney U-test. Will perform these tests adjusting for 6 pairwise multiple comparisons among the four groups using the Bonferroni?s correction method.
Adherence as measured by frequency of 6-MP dosing as a continuous variable using MEMS? defined as the number of days the MEMS? Cap openings are recorded, taken as a percentage of days doses were prescribed during the study period | Up to 169 days
  Will initially perform an exploratory data analysis on distributions across the four groups using side-by-side boxplots, histograms, and summary quantities (mean, median, quartiles, standard deviations, inter-quartile-range, etc.). If central values summarize across-group differences well, then mean and median of the distribution will be compared between 6 pairs of the four ethnic groups using the two-sample t-test and the Mann-Whitney U-test. Will perform these tests adjusting for 6 pairwise multiple comparisons among the four groups using the Bonferroni?s correction method.
Self-report of adherence to 6-MP by questionnaire, defined as the number of days doses of 6-MP are reported to being taken, as a percentage of days doses were prescribed during the study period | 169 days
  Will initially perform an exploratory data analysis on distributions across the four groups using side-by-side boxplots, histograms, and summary quantities (mean, median, quartiles, standard deviations, inter-quartile-range, etc.). If central values summarize across-group differences well, then mean and median of the distribution will be compared between 6 pairs of the four ethnic groups using the two-sample t-test and the Mann-Whitney U-test. Will perform these tests adjusting for 6 pairwise multiple comparisons among the four groups using the Bonferroni?s correction method.
EFS | Up to 10 years
  For each of the three types of adherence measures, will fit independent Cox?s proportional-hazard models to assess the prognostic significance of the adherence measure on EFS, after adjusting for known predictors of disease outcome, including the National Cancer Institute risk group (based on the age at diagnosis and presenting white cell count) and chromosomal abnormalities.
Critical level of adherence (measured independently by 6TGN/MethylTIMP, MEMS?, self-report) that has a significant impact on EFS | Up to 10 years
  Will fit a separate Cox regression model to each of the three adherence measures (i.e., 6TGN, MeTIMP, MEMS, and self-report). Using no more than several knots, the natural spline (a special type of cubic splines) fits a very wide range of smoothly changing adherence effects. The adherence effects on EFS will be visualized graphically. This will be the primary approach for defining the critical level of adherence. To confirm the spline analysis results, will categorize the continuous adherence measures into multiple levels and estimate the effect of each adherence level.
Prevalence of adherence to 6-MP by ethnicity (measured independently by 6TGN/MethylTIMP, MEMS?, Self-report) that has a significant impact on EFS | Up to 10 years
  Will describe the prevalence of non-adherence by race/ethnicity and compare the prevalence by using two-tailed chi-squared test (with a Yates' correction).
Behavioral, socio-demographic predictors of adherence using the questionnaire data | Up to 10 years
  The reasons for non-adherence will be assessed. The relationship between adherence to 6-MP as reported by the patients/parents and the independent behavioral variables knowledge of medications, understanding of treatment regimen, extent of treatment side effects, length of treatment, and beliefs about the efficacy of the regimen, beliefs and attitudes towards health and medical care will be evaluated descriptively first using standard parametric or non-parametric tests, and then analytically by logistic regression (dichotomous adherence) or linear regression (continuous adherence).
Pill-taking practices using the MEMS? data | Up to 169 days
  Using the MEMS? output data, the adherence report will be analyzed for: i) longest and shortest interval between doses in hours; ii) percent prescribed doses taken, and iii) percent prescribed doses taken on schedule.
Impact of adherence (measured independently by 6TGN/MethylTIMP, MEMS, self-report) on ethnic/racial differences in EFS | Up to 10 years
  Will fit independent Cox?s proportional-hazard models to assess the impact of adherence measure on EFS, after adjusting for known predictors of disease outcome, including the National Cancer Institute risk group (based on the age at diagnosis and presenting white cell count) and chromosomal abnormalities.

SECONDARY OUTCOMES:
Concordance among red cell thiopurine metabolite levels, electronic pill monitoring, and self-reported adherence among the ethnic/racial groups | Up to 168 days
  Correlations between mean dosage- and TPMT-normalized serial red cell 6-MP metabolites and mean adherence by electronic pill monitoring system and self-report will be assessed for statistical significance by Spearman's rank correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Bhatia, Principal Investigator — Children's Oncology Group
Locations (135):
- United States (124):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Brooklyn Hospital Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Victoria Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Wadhwa A, Chen Y, Hageman L, Hoppmann A, Angiolillo A, Dickens DS, Neglia JP, Ravindranath Y, Ritchey AK, Termuhlen A, Wong FL, Landier W, Bhatia S. Poverty and relapse risk in children with acute lymphoblastic leukemia: a Children's Oncology Group study AALL03N1 report. Blood. 2023 Jul 20;142(3):221-229. doi: 10.1182/blood.2023019631. PMID 37070673
- [Derived] Yang JJ, Landier W, Yang W, Liu C, Hageman L, Cheng C, Pei D, Chen Y, Crews KR, Kornegay N, Wong FL, Evans WE, Pui CH, Bhatia S, Relling MV. Inherited NUDT15 variant is a genetic determinant of mercaptopurine intolerance in children with acute lymphoblastic leukemia. J Clin Oncol. 2015 Apr 10;33(11):1235-42. doi: 10.1200/JCO.2014.59.4671. Epub 2015 Jan 26. PMID 25624441
- [Derived] Bhatia S, Landier W, Hageman L, Kim H, Chen Y, Crews KR, Evans WE, Bostrom B, Casillas J, Dickens DS, Maloney KW, Neglia JP, Ravindranath Y, Ritchey AK, Wong FL, Relling MV. 6MP adherence in a multiracial cohort of children with acute lymphoblastic leukemia: a Children's Oncology Group study. Blood. 2014 Oct 9;124(15):2345-53. doi: 10.1182/blood-2014-01-552166. Epub 2014 May 14. PMID 24829202